CLINICAL TRIAL: NCT00716690
Title: Enhancement of Hematopoietic Stem Cell Engraftment by Multi Donor Stem Cell Transplantation (MDT) From 2 Mismatched Donors, a Phase I-II Open Study
Brief Title: Multi Donor Mismatched Stem Cell Transplantation (MDT)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, SHAPIRA MICHAEL, Prof Shapira, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYS-04-HMO-CTIL
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Graft-Versus-Host Disease
Keywords: Stem cell transplantation; GVHD
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental)
  Interventions: Procedure: Multi donor stem cell transplantation

INTERVENTIONS:
Procedure: Multi donor stem cell transplantation — stem cell transplantation from 2 donors

SUMMARY:
The proposed research focuses on the development of innovative protocol of mismatched stem cell transplantation with combined 2 different haplo stem cell transplantation (SCT) donors which are mismatched to the recipient (and preferably to each other), in a patient in need for SCT, lacking an HLA match related or an unrelated donor. This innovative protocol named multi donor stem cell transplantation (MDT) is designed to facilitate engraftment even when reduced intensity conditioning or a low cell dose are used, improve the graft vs. leukemia (GVL) effect and enhance immune reconstitution (using quantitative and qualitative parameters).

ELIGIBILITY:
Inclusion criteria:

1. Patient age 0-70 years old with leukemia in 1st remission at high risk of relapse because of unfavorable prognostic features, at 2nd CR or MDS without an readily available matched donor (related or unrelated).
2. Patients must have a mismatched donor willing and capable of donating peripheral blood stem cells and/or bone marrow progenitor cells using conventional techniques, and lymphocytes if indicated (mismatched defined as 3/6-4/6 HLA matching).
3. Each patient / patient's guardian must sign written informed consent.
4. Patients must have an ECOG PS ≤ 2; Creatinine <2.0 mg/dl; Ejection fraction >40%; DLCO >50% of predicted; Serum bilirubin <3 gm/dl; elevated GPT or GOT <3 x normal values.

Exclusion criteria:

1. Not fulfilling any of the inclusion criteria.
2. Not in CR (if the indication for transplant is leukemia).
3. Active life-threatening infection.
4. Overt untreated infection.
5. HIV seropositivity, Hepatitis B or C antigen positivity with evidence of active hepatitis.
6. Pregnant or lactating women.
7. Donor contraindication (HIV seropositive confirmed by Western Blot, Hepatitis B antigenemia, HCV, evidence of bone marrow disease, unable to donate bone marrow or peripheral blood due to concurrent medical condition).
8. Previous autologous or allogeneic stem cell transplantation.
9. Inability to comply with study requirements.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-07; Primary Completion 2020-01 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Day of neutrophil engraftment | 30d
Day of platelet engraftment>20x10(9)L | 30
Acute GVHD occurrence>2 | 100d
Disease free survival | 100d

SECONDARY OUTCOMES:
Day of platelet engraftment>50x10(9)/L | 30d
Time of acute GVHD | 100d
GVHD grade | 100d
Overall survival | 100 days
Infections incidence | 100d
transplant-related mortality | 100d
Transplant related toxicity | 100d
Immune reconstitution | 100d

CONTACTS AND LOCATIONS:
Overall Officials: Michael Y Shapira, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel